CLINICAL TRIAL: NCT02398396
Title: Investigating Meningococcal Vaccines in Adults - An Exploratory, Open-label, Immunogenicity Study of a Licensed Meningococcal Capsular Group B Vaccine (4CMenB, Bexsero®) in Adults
Brief Title: Investigating Meningococcal Vaccines in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OVG 2014/12
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2018-10

CONDITIONS: Meningococcal Vaccines; Meningococcal Infections; Neisseria Meningitidis; Factor H-binding Protein, Neisseria Meningitidi
MeSH Terms: conditions — Meningococcal Infections | interventions — 4CMenB vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label: 4CMenB (Bexsero®) (Experimental)
  Interventions: Biological: 4CMenB (Bexsero®) - Novartis Vaccines and Diagnostics

INTERVENTIONS:
Biological: 4CMenB (Bexsero®) - Novartis Vaccines and Diagnostics — 4CMenB vaccine (Bexsero - Novartis Vaccines and Diagnostics) 0.5ml intra-muscularly; two doses, administered 2 months apart. Each dose of vaccine contains recombinant Neisseria meningitidis group B NHBA fusion protein (50 micrograms); recombinant Neisseria meningitidis group B NadA protein (50 micrograms); recombinant Neisseria meningitidis group B FHbp fusion protein (50 micrograms) and Outer membrane vesicles (OMV) from Neisseria meningitidis group B strain NZ98/254 (25 micrograms measured as amount of total protein containing the PorA P1.4)

SUMMARY:
This study will be an open label, exploratory immunogenicity study conducted by the Oxford Vaccine Group, University of Oxford. This study will investigate the breadth of protective activity of serum anti-FHbp antibody responses of adults immunized with 4CMenB (Bexsero®) vaccine as well as investigating the nature of the B-cell and T-cell responses induced by vaccination.

The investigators aim to enroll 15 to 20 healthy adults aged 18 to 60, who will be immunized with two doses of 4CMenB (Bexsero®) two months apart according to the licensed schedule. Blood samples will be obtained at baseline and after each dose of vaccine.

DETAILED DESCRIPTION:
Neisseria meningitidis (N. meningitidis, meningococcus) is a leading cause of bacterial meningitis and septicaemia worldwide. The introduction of serotype specific glycoconjugate vaccines into the routine infant immunization schedule, in countries such as the United Kingdom, has led to dramatic reductions in the burden of disease. The development of effective vaccines against capsular group B N. meningitidis has long been an unmet need and has necessitated the development of novel approaches to vaccine design. In 2013, the first capsular group B meningococcal vaccine was licensed in the UK. The new vaccine (4CMenB, trade name Bexsero ®), is manufactured by Novartis Vaccines and contains four components - a recombinant Factor H binding protein (FHbp), Neisseria meningitidis capsular group B Neisseria Heparin Binding Antigen (NHBA) fusion protein, recombinant Neisseria meningitidis group B Neisserial adhesin A (NadA) protein and Outer membrane vesicles (OMV) from Neisseria meningitidis group B strain NZ98/254 containing PorA P1.4. This multicomponent vaccine is also referred to as the "four component meningococcal B" or "4CMenB" vaccine.

Factor H binding protein is an important virulence factor expressed on the surface of N. meningitidis and is a key component of the 4CMenB vaccine. It has been established that the function of FHbp is to bind human complement factor H, whose physiological function in turn is to act as an important down-regulator of the host alternative complement pathway. Binding of human factor H to the bacterial surface via FHbp is thought to interfere with complement mediated lysis and is an important immune evasion strategy of N. meningitidis. Consequently, FHbp is a logical target for a protective vaccine against capsular group B N. meningitidis.

There remain several gaps in our knowledge about the underlying mechanisms by which human antibodies to FHbp elicit complement mediated bactericidal activity. In humans immunised with vaccines containing FHbp, the antigen (FHbp) is expected to form a complex with human factor H. The precise epitopes targeted by anti-FHbp antibodies in vaccinees have not been fully elucidated. Conceivably, the formation of a FHbp-factor H complex following vaccination may prevent the exposure of key FHbp epitopes. Therefore, it is not known whether the interaction between FHbp and human Factor H affects the bactericidal activity of antibodies produced following vaccination with 4CMenB.

This study will investigate the breadth of protective activity of serum anti-FHbp antibody responses of adults immunized with 4CMenB (Bexsero®) vaccine as well as investigating the nature of the B-cell and T-cell responses induced by vaccination.

We aim to enroll 15 to 20 healthy adults aged 18 to 60, who will be immunized with two doses of 4CMenB (Bexsero®) two months apart according to the licensed schedule. Sera will be obtained at baseline and after each dose of vaccine, which will be assayed for IgG antibody responses to FHbp by ELISA, as well as for bactericidal activity against a panel of genetically diverse meningococcal strains and for the ability to inhibit binding of FH to FHbp. Other assays for meningococcal immunity may also be performed such as antibody binding to live bacteria measured by flow cytometry, and the ability of the serum antibodies to confer passive protection in an infant rat bacteraemia model. Laboratory analyses to quantify the B- and T-cell responses specific to the 4CMenB vaccine will be performed using peripheral blood mononuclear cells (PBMCs) derived from study participants sampled before, and after each dose. We will also explore whether the formation of the FH-FHbp complex results in the generation of cross-reactive antibodies directed against Factor H.

This will be the first study in humans to explore in detail the anti-FHbp characteristics generated following immunization with 4CMenB (Bexsero®) and offers a unique opportunity to use a licensed vaccine to improve our understanding of how to induce efficient protective responses. It is hoped that the results obtained from this study will contribute to our understanding of the host response to vaccination against capsular group B N. meningitidis.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years to 60 years inclusive on the day of first vaccination.
* To be in good health as determined by medical history, physical examination and clinical judgment of the investigators.
* Agree (in the Investigator's opinion) to comply with all study requirements
* Agree to allow his or her General Practitioner (and/or Consultant if appropriate), to be notified of participation in the study
* Agree to provide their National Insurance/Passport number for the purposes of TOPS registration and bank account information for the purpose of reimbursement for the duration of their participation.

Exclusion Criteria:

* Have any known or suspected impairment or alteration of immune function, resulting from, for example:

  * Congenital or acquired immunodeficiency (including IgA deficiency)
  * Human Immunodeficiency Virus (HIV) infection or symptoms/signs suggestive of an HIV-associated condition
  * Autoimmune disease
  * Receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 12 months or long-term systemic corticosteroid therapy.
  * Chronic illness that could interfere with immunological function or donation of the required volumes of blood (e.g. cardiac or renal disease, diabetes, or auto-immune disorders).
* Receipt of a live vaccine within 4 weeks prior to vaccination or a killed vaccine within 7 days prior to vaccination.
* History of group B meningococcal vaccination
* Have received a dose of a meningococcal groups A, C, W, Y conjugate vaccine within 30 days of enrolment or wish to receive a dose of this vaccine during the study period.
* Plan to receive any vaccine other than the study vaccine within 4 weeks following vaccination.
* History of severe allergic reaction after vaccination or known hypersensitivity to any vaccine component
* History of meningococcal disease
* Receipt of blood, blood products, or plasma derivatives within the past 3 months.
* Recent significant blood donation (e.g., to the National Blood Service) within 8 weeks of enrolment, or plans to donate blood during the study period.
* Thrombocytopenia or any bleeding disorder.
* Pregnancy as confirmed by a positive pregnancy test, or currently breastfeeding.
* Enrolled in another study, which, in the opinion of the investigator, could compromise the integrity of either study being conducted.
* A member of staff on the delegation log
* According to the TOPS database, have recently taken part in a significant number of other studies, which, in the opinion of the investigator, warrant exclusion from further studies.
* Have any condition, which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
To characterise the breadth of protective activity of serum anti-FHbp antibody responses of adults immunised with 4CMenB (Bexsero) vaccine | 3 months
  As measured by IgG antibody responses to FHbp as measured by serum bactericidal activity against a panel of genetically diverse meningococcal strains

SECONDARY OUTCOMES:
To investigate the nature of the B-cell response that supports the induction of antibody with functional activity following vaccination with 4CMenB | 3 months
  Quantification of circulating vaccine-induced memory B-cells specific for vaccine antigens before and after each, dose.
To investigate the nature of the T-cell response that supports the induction of antibody with functional activity following vaccination with 4CMenB | 3 months
  Quantification of vaccine-induced, antigen specific T-cell responses and associated cytokine production before and after each dose.
Determine whether adults immunised with 4CMenB develop serum IgG and IgM antibodies to human FH | 3 months
  Serum IgG and IgM antibodies to human FH will as measured by ELISA

OTHER OUTCOMES:
Exploratory immunology to investigate the role of anti-FHBp antibodies in meningococcal immunity | 3 months
  Exploratory assays including Factor H (FH) - FHbp binding inhibition assays, antibody binding to live bacteria measured by flow cytometry, passive transfer experiments using infant rat bacteraemia model.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Giuntini S, Lujan E, Gibani MM, Dold C, Rollier CS, Pollard AJ, Granoff DM. Serum Bactericidal Antibody Responses of Adults Immunized with the MenB-4C Vaccine against Genetically Diverse Serogroup B Meningococci. Clin Vaccine Immunol. 2017 Jan 5;24(1):e00430-16. doi: 10.1128/CVI.00430-16. Print 2017 Jan. PMID 27847367